CLINICAL TRIAL: NCT06828289
Title: Observational Study of Rivastigmine Mini-Tablet in Patients with Alzheimer's Disease
Brief Title: Rivastigmine Mini-Tablet for Alzheimer's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KBLT
Record Dates: First submitted 2025-02-11; First posted 2025-02-14 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Rivastigmine Mini-Tablet: Start with a dose of 1.5 mg twice daily (bid), titrate every two weeks, and the maximum dose should not exceed 12 mg.
  Interventions: Drug: Rivastigmine Mini-Tablet
- Donepezil Hydrochloride: Start with 5mg taken once daily before bedtime. If the patient tolerates the initial dose well, it will be increased to 10 mg per day after four weeks.
  Interventions: Drug: Donepezil Hydrochloride

INTERVENTIONS:
Drug: Rivastigmine Mini-Tablet — Treatment group: Rivastigmine Mini-Tablet
  Groups: Rivastigmine Mini-Tablet
Drug: Donepezil Hydrochloride — Control group: Donepezil Hydrochloride
  Groups: Donepezil Hydrochloride

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of rivastigmine mini-tablets in individuals diagnosed with mild to moderate Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Rivastigmine has received approval for the treatment of Alzheimer's disease. The rivastigmine mini-tablet represents an innovative drug formulation designed to address swallowing difficulties by reducing the size of the dosage form, while also minimizing gastrointestinal side effects through an optimized drug release mechanism. This multi-center, observational study aims to evaluate the effectiveness, safety, and patient compliance associated with rivastigmine mini-tablets in individuals diagnosed with Alzheimer's disease. Assessments will be conducted at the 3rd, 6th, and 12th months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older
* Meet the National Institute of Aging-Alzheimer's Association clinical criteria for probable Alzheimer's disease
* Have a Mini-Mental State Examination score of 10 to 24 at Screening and Baseline
* Geriatric Depression Scale score <=7 at Screening
* Hachinski Ischemic Scale <=4 at Screening
* Brain MRI should meet: no infarcts in key areas (thalamus, hippocampus, entorhinal cortex, perirhinal cortex, angular gyrus, etc.), ≤ 2 stroke lesions > 1.5 cm in diameter, and Fazekas Scale - assessed white matter lesion grade

  * 2.
* Patients whose caregivers are well-informed about the patients' condition and, if possible, live with them.
* Provide written informed consent

Exclusion Criteria:

* Any systemic or neurological condition that could contribute to cognitive impairment above and beyond that caused by the participant's Alzheimer's disease
* Any psychiatric diagnosis or symptoms (hallucinations, major depression, delusions, etc) interfering with study procedures
* An advanced, severe or unstable disease of any type (cardiac, respiratory, gastrointestinal, renal disease, etc) that may interfere with efficacy evaluations
* Subjects treated with medication for dementia two weeks prior to baseline

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Alzheimer's disease
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in Clinical Dementia Rating Sum of Boxes (CDR-SB) | Baseline to 12 months
  CDR-SB range 0-18, with higher scores indicating more severe dementia.

SECONDARY OUTCOMES:
Changes from baseline in Mini-Mental State Examination (MMSE) scale scores | Baseline to 12 months
  MMSE range 0-30, with higher scores indicating better cognitve functioning.
Changes from baseline in Neuropsychiatric Inventory (NPI) scale scores | Baseline to 12 months
  NPI score range is 0-144 for patient assessment and 0-60 for caregiver distress assessment. In patient assessment, higher scores indicate more severe neuropsychiatric disorders; in caregiver distress assessment, higher scores indicate greater distress.
Changes from baseline in Alzheimer's Disease Cooperative Study ADL（ADCS-ADL)） scores | Baseline to 12 months
  ADCS-ADL range 0-78, with higher scores indicating better functional ability in daily activities.
Concentration Changes from Baseline of Plasma Biomarkers (Aβ42/40, p - tau181, p - tau217, NfL and GFAP） | Baseline to 12 months
  The plasma biomarkers include Aβ42/40，p-tau181, p-tau217, NfL and GFAP.
Safety and Tolerability | Baseline to 12 months
  The adverse event, discontinuation due to intolerability, etc will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Yongan Sun, Phd, Principal Investigator — Peking University First Hospital